CLINICAL TRIAL: NCT03365219
Title: Alexis O-Ring Wound Retractor for the Prevention of Post-cesarean Surgical Site Infections: A Randomized Controlled Trial
Brief Title: Alexis O-Ring Wound Retractor for the Prevention of Post-cesarean Surgical Site Infections
Acronym: Alexis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-188
Record Dates: First submitted 2015-06-09; First posted 2017-12-07 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-05

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Site Infection; Cesarean delivery infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alexis Retractor (Experimental): This group received an Alexis O-Ring Wound Retractor during cesarean delivery.
  Interventions: Device: Alexis O-Ring Wound Retractor
- Standard Surgical Retractors (Active Comparator): This group received routine hand-held metal retractors as needed by the surgical team during cesarean delivery.
  Interventions: Other: Standard Surgical Retractors

INTERVENTIONS:
Device: Alexis O-Ring Wound Retractor — A flexible self-retaining plastic Alexis retractor was used in place of standard surgical retractors.
  Arms: Alexis Retractor
Other: Standard Surgical Retractors — Routine hand-held metal retractors as needed by the surgical team
  Arms: Standard Surgical Retractors

SUMMARY:
Post cesarean section surgical site infection (SSI) is a common complication that can affect patient recovery and overall outcome. Several approaches have been studied to improve SSI rates such as timing of antibiotic administration and skin preparation. Alexis retractors have been suggested as a reasonable option to decrease SSI. However, to date there is only one randomized controlled study assessing its efficacy. The aim of this study is to whether Alexis wound retractors are beneficial in preventing cesarean section SSI.

DETAILED DESCRIPTION:
The study design was a randomized controlled study to evaluate wound infection rates in patients undergoing a cesarean delivery. The patients were randomized into two sub- groups; the first group received routine hand-held metal retractors as needed by the surgical team, and the second group received an Alexis Wound Retractor. Inclusion criteria included: maternal age of at least 18 years, a gestational age of at least 24 0/7 wks by best obstetric estimate, a viable gestation, a non-emergent cesarean delivery, and a planned transverse skin incision. Deliveries included: primary cesarean for failed induction, maternal request, or other obstetric indications; and repeat cesarean deliveries that were elective or had obstetric indications (such as spontaneous labor in a subject with a term gestation and with history of 2 or more prior cesarean deliveries). Exclusion criteria included chorioamnionitis, chronic corticosteroid therapy, a prior abdominal vertical skin incision scar or planned vertical incision, history of a prior wound infection or separation, a planned cesarean hysterectomy, or maternal or fetal complications requiring an emergent delivery.

Randomization was done using a web-based randomization generator. Variables were allocated as: 1 for Alexis, and 0 for conventional surgical retractors. Packages including consent forms, data sheets, and the randomized allocation were prepared for the entire study and were stored in one office. Study packets were prepared to include a sealed envelope indicating randomization to be opened after the consent form was signed. Only after randomization, the Alexis retractor was opened and placed on the surgical field.

Prior to initiation of the study, in-service sessions were conducted with OB surgical teams to facilitate the use of the retractors. Information provided included optimal use of the retractor and selection of the appropriate retractor size. The primary surgeon of each case was previously trained by the principle investigator in placement of the retractor on actual patients.

Once a decision was made to proceed with cesarean delivery, the subject was approached and offered to participate in the study. After the patient had been enrolled and consent forms signed, an allocated envelope for each study subject determined which arm of the study to which the patient would be randomized; no other management decisions was made as part of the RCT. Surgical decisions were independent of the patient's designated study arm and retractor type. Such decisions included: type of anesthesia, length of transverse skin incision , method of tissue dissection (blunt vs. instrumental), creation of bladder flap, size and nature of uterine incision (transverse, low vertical, classical, J-type, T-incision), surgical material used, exteriorization of the uterus, manual vs. spontaneous delivery of placenta, layer closure techniques (bladder flap, peritoneum, subcutaneous tissue), and skin closure technique (staples, subcuticular sutures). Skin preoperative preparation was performed as standard with ChloraPrep® Applicator (2% Chlorhexidine gluconate and 70% isopropyl alcohol). Intravenous antibiotics were given preoperatively in accordance to national guidelines (12). The primary outcome of this study was the development of a surgical site infection after cesarean delivery within two weeks after cesarean.

Incisions were checked daily in-house. However, the exams that were used in this study to determine the occurrences of SSI were the first exam done in the outpatient setting for removal of staples (post op days 5 - 7), and the two week post partum visit (post op days 14 - 18). SSIs were diagnosed according to the Centers for Disease Control and Prevention (CDC) criteria.(13). The most commonly seen characteristics were purulent drainage or localized swelling and/or redness of the surgical wound.

In addition, other wound complications were also assessed and included: seroma (wounds with clear drainage) and/or hematomas. Other secondary outcomes included skin time to uterine incision (minutes) , exteriorization of the uterus(yes, no), total operative time (minutes), estimated blood loss (mL) estimated by the primary surgeon, and postoperative pain based on a subjective 1-10 pain scale, assessed 4 times daily while hospitalized and at the outpatient visits previously mentioned.

An initial sample size estimate was performed using the frequentist approach with an assumption of power 80% and Type 1 error = 5% (2-sided). The primary outcome of the study is expected to occur in 15% of women in the "usual care" group. In order to detect a 50% reduction (15% to 7.5%) in the rate of wound complications with the use of the Alexis retractor, a total sample size of 564 women will be needed (282 per group). The planned study was to be carried out at two distinct sites: the University of Texas Medical Branch in Galveston (UTMB) and the University of Texas in Houston. The Institutional Review Board of UTMB-Galveston IRB # 10-188 approved the study.

ELIGIBILITY:
Inclusion Criteria:

* maternal age of at least 18 years
* a gestational age of at least 24 0/7 wks by best obstetric estimate
* a viable gestation
* a non-emergent cesarean delivery
* a planned transverse skin incision
* Deliveries included: primary cesarean for failed induction, maternal request, or other obstetric indications; and repeat cesarean deliveries that were elective or had obstetric indications (such as spontaneous labor in a subject with a term gestation and with history of 2 or more prior cesarean deliveries)

Exclusion Criteria:

* chorioamnionitis
* chronic corticosteroid therapy
* prior abdominal vertical skin incision scar or planned vertical incision
* history of a prior wound infection or separation
* planned cesarean hysterectomy
* maternal or fetal complications requiring an emergent delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | Time of surgery up to 14 post operative days
  Assessed as present or absent. Defined as the development of wound infection, seroma, or other wound disruption in patients who underwent a cesarean delivery

SECONDARY OUTCOMES:
Postoperative pain | Time of surgery up to 14 post operative days
  Patients are asked to report pain on a scale of 1-10, 1 no pain and 10 the worst pain.
Estimated blood loss | intraoperative assessment
  Defined as the amount of blood loss during the cesarean delivery as estimated by the operating surgeons.
Uterus exteriorization | intraoperative assessment
  Quantified as yes or no; defined as whether or not the surgeons' exteriorized the uterus extra-corporally (removed from abdominal cavity) at any time of the cesarean delivery
Total operative time | intraoperative assessment
  Defined as the total length of time in minutes required to perform the cesarean delivery from time of initial skin incision to completion of skin closure.

OTHER OUTCOMES:
Apgar scores | Assessed in every infant at 1 minute and 5 minutes of life
  Score given by pediatrician or pediatric provider to each infant at 1 and 5 minutes of life
Gestational age at time of delivery | at time of delivery
  Completed gestational age in weeks
Infant weight | At time of delivery
  Infant Weight in kg
Type of gestation | Noted at the time of delivery
  Singleton or multiple fetus
Maternal hypertension | At the time of delivery until 14 days after delivery
  Systolic blood pressure greater than 140 and diastolic blood pressure greater than 90 mmHG

CONTACTS AND LOCATIONS:
Overall Officials: Gayle L Olson, MD, Principal Investigator — University of Texas Medical Branch in Galveston; George Saade, MD, Study Chair — University of Texas Medical Branch in Galveston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menacker F, Hamilton BE. Recent trends in cesarean delivery in the United States. NCHS Data Brief. 2010 Mar;(35):1-8. PMID 20334736
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Stone PW, Braccia D, Larson E. Systematic review of economic analyses of health care-associated infections. Am J Infect Control. 2005 Nov;33(9):501-9. doi: 10.1016/j.ajic.2005.04.246. PMID 16260325
- [Background] Moir-Bussy B, Hutton R, Thompson J. Wound infection after caesarean section. Nurs Times. 1985 Jun 5-11;81(23):suppl 13-4. No abstract available. PMID 3847906
- [Background] Rauk PN. Educational intervention, revised instrument sterilization methods, and comprehensive preoperative skin preparation protocol reduce cesarean section surgical site infections. Am J Infect Control. 2010 May;38(4):319-23. doi: 10.1016/j.ajic.2009.10.004. Epub 2010 Feb 19. PMID 20171756
- [Background] Schneid-Kofman N, Sheiner E, Levy A, Holcberg G. Risk factors for wound infection following cesarean deliveries. Int J Gynaecol Obstet. 2005 Jul;90(1):10-5. doi: 10.1016/j.ijgo.2005.03.020. PMID 15913620
- [Background] Tran TS, Jamulitrat S, Chongsuvivatwong V, Geater A. Risk factors for postcesarean surgical site infection. Obstet Gynecol. 2000 Mar;95(3):367-71. doi: 10.1016/s0029-7844(99)00540-2. PMID 10711546
- [Background] Weiss JL, Malone FD, Emig D, Ball RH, Nyberg DA, Comstock CH, Saade G, Eddleman K, Carter SM, Craigo SD, Carr SR, D'Alton ME; FASTER Research Consortium. Obesity, obstetric complications and cesarean delivery rate--a population-based screening study. Am J Obstet Gynecol. 2004 Apr;190(4):1091-7. doi: 10.1016/j.ajog.2003.09.058. PMID 15118648
- [Background] Cedergren MI. Maternal morbid obesity and the risk of adverse pregnancy outcome. Obstet Gynecol. 2004 Feb;103(2):219-24. doi: 10.1097/01.AOG.0000107291.46159.00. PMID 14754687
- [Background] ACOG Practice Bulletin No. 120: Use of prophylactic antibiotics in labor and delivery. Obstet Gynecol. 2011 Jun;117(6):1472-1483. doi: 10.1097/AOG.0b013e3182238c31. No abstract available. PMID 21606770
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Result] Cheng KP, Roslani AC, Sehha N, Kueh JH, Law CW, Chong HY, Arumugam K. ALEXIS O-Ring wound retractor vs conventional wound protection for the prevention of surgical site infections in colorectal resections(1). Colorectal Dis. 2012 Jun;14(6):e346-51. doi: 10.1111/j.1463-1318.2012.02943.x. PMID 22568647